CLINICAL TRIAL: NCT06462274
Title: Biomarkers and Imaging Markers Screening for Intracerebral Hemorrhage Patients
Brief Title: Biomarkers and Imaging Markers for ICH
Status: Recruiting | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Rong Hu, MD, Associate professor, Associate chief neurosurgeon, Southwest Hospital, China
Other Study IDs: Neurosurg03
Record Dates: First submitted 2016-01-31; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Central laboratory biobank
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ICH group: Patients with CT-demonstrated Intracerebral Hemorrhage (ICH) within 72 hours after symptom onset admitted to Southwest hospital.
  Interventions: Other: body sample collection and imaging scan
- Control group: Age- and sex-matched healthy individuals were recruited from volunteers.
  Interventions: Other: body sample collection and imaging scan

INTERVENTIONS:
Other: body sample collection and imaging scan

SUMMARY:
Intracerebral hemorrhage (ICH) is a subtype of stroke associated with high mortality and disability. Basic and clinical research has contributed to our understanding of the complex pathophysiology in ICH. However, questions regarding acute diagnosis, therapeutic decisions, and prognostication of ICH remain unanswered. Molecular biomarkers and imaging markers have revolutionalized diagnosis and treatment of many diseases, such as troponin use in myocardial infarction and magnetic resonance imaging (MRI) scan in ischemic stroke. Therefore, the investigators aim to discovery the potential biomarkers by screening samples of blood, cerebral spinal fluid, urine, saliva, and even tissues (if available) from ICH patients, and imaging markers via serial multimodality imaging scans such as computed tomography(CT), magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), positron emission tomography (PET), etc. These molecular and imaging markers would assist in contributing additional information to current tools for onset warning, diagnosis, therapy monitoring, risk stratification, intervention and prognosis for ICH patients.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is one of the most serious subtypes of stroke, affecting approximately 2-3 million people worldwide each year. About one third of people with ICH die early after onset and the majority of survivors are left with major long-term disability. Today little is known about the characteristic changes in molecules from body samples and pictures from multimodality imaging scans. In this study, the investigators aim to reveal the potential biomarkers by screening samples of blood, cerebral spinal fluid, urine, saliva, and even tissues (if available) from ICH patients, and imaging markers via serial multimodality imaging scans such as computed tomography(CT), magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), positron emission tomography (PET), etc, which will bring insights into pathophysiological mechanisms and addition of new tools for onset warning, diagnosis, therapy monitoring, risk stratification, intervention and prognosis for ICH patients.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-80 years
2. Hematoma size is more than 5 ml
3. Evidence of a spontaneous ICH on CT scan
4. Patient within 72 hours of ictus
5. Glasgow Coma Scale (GCS) Score of 5-15.
6. The history of hypertension

Exclusion Criteria:

1. Individuals with age < 18 years or > 80 years
2. Clear evidence that the hemorrhage is due to an aneurysm, arteriovenous malformation or other cerebrovascular diseases.
3. ICH secondary to tumor or trauma..
4. If the haematological effects of any previous anticoagulants are not completely reversed.
5. Patients with heart insufficiency, lungs insufficiency, renal insufficiency, hepatic insufficiency, autoimmune diseases and other organ diseases with severe dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Individuals aged 18-80 years
  2. Evidence of a spontaneous ICH on CT scan
  3. Patient within 72 hours of ictus
  4. Glasgow Coma Scale (GCS) Score of 5-15.
  5. The history of hypertension
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01-01; Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers | Immediately after collecting tissues
  Diseased tissue from the patient is collected at the time of hematoma removal. These tissues are then immediately prepared and detected by proteome mass spectrometry. The results will be further analyzed by bioinformatics analysis to reveal the expression of proteins in the diseased tissues of patients with intracerebral hemorrhage as potential biomarkers.
CT imaging features | Within 1 month of onset
  Patients will undergo CT imaging examinations to evaluate the patient's hematoma volume, hematoma location, hematoma morphology, hematoma density and other imaging characteristics
CTA imaging markers | Within 1 month of onset
  The patient will undergo CTA imaging to evaluate the cerebrovascular features of the patient
MR imaging markers | Within 1 month of onset
  Magnetic resonance imaging was performed to evaluate the patient's hematoma morphology, signal, and edema around the hematoma cavity

SECONDARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) | 1 year
  GOS-E subdivides the categories of severe and moderate disability and good recovery using a scale of 1 to 8 where 1 = death, 2 = vegetative state, 3 = lower severe disability, 4 = upper severe disability, 5 = lower moderate disability, 6 = upper moderate disability, 7 = lower good recovery, and 8 = upper good recovery. Structured telephone interviews have been developed and validated for the GOS-E and these questions were incorporated into the follow-up survey. GOS-E was dichotomized into unfavorable (1 to 4) and favorable (5 to 8) outcomes.
modified Rankin scale (mRS) | 1 year
  Functional outcome (comparing the intervention group to the control), assessed with the modified Rankin Scale (mRS) at 6 months.The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Hu, Ph.D, Principal Investigator — Southwest Hospital, China
Locations (1):
- Department of Neurosurgery , Southwest Hospital, Third Military Medical University,, Chongqing, Chongqing Municipality, China